CLINICAL TRIAL: NCT05139368
Title: RT-PACE: A Pilot Study of Adjuvant Hypo-Fractionated Radiotherapy for Non-Metastatic Cervical and Endometrial Cancer
Brief Title: Hypofractionated Radiotherapy for the Treatment of Cervical or Endometrial Cancer
Acronym: RT-PACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI144462; NCI-2021-12258 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI144462 (Other: Huntsman Cancer Institute/University of Utah); P30CA042014 (NIH)
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cervical Carcinoma; Endometrial Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Radiation Dose Hypofractionation; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (hypo-fractionated radiotherapy) (Experimental): Patients undergo hypo-fractionated radiotherapy over 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated

SUMMARY:
This clinical trial studies the feasibility of using hypo-fractionated radiotherapy for the treatment of cervical or endometrial cancer. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the trial as feasible and to assess the impact upon acute gastrointestinal toxicity in the third week of pelvic radiotherapy following a hypo-fractionated schedule.

SECODARY OBJECTIVES:

I. To estimate impact upon acute urinary toxicity. II. To estimate impact upon patient reported gastrointestional toxicity. III. To assess acute quality of life following treatment. IV. To quantify acute financial toxicity following treatment. V. To assess satisfaction with decision-making following treatment. VI. To assess the overall survival throughout 3 years of post-treatment follow-up.

OUTLINE:

Patients undergo hypo-fractionated radiotherapy over 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1, 3, and 6 months and then at 1, 2, and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged >= 18 years
* Pathologically confirmed malignancy of the cervix or endometrium. Non-epithelial histologies are permitted. Adenocarcinoma in situ is also permitted
* Patients must be status post hysterectomy for initial management of cervix or endometrial cancer
* Subject must have non-metastatic disease as determined by clinical exam or computed tomography (CT) or positron emission tomography (PET)/CT imaging
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 from toxicities related to any prior cancer therapy, unless considered clinically not significant by the treating investigator
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines
* Life expectancy of > 2 years
* Chemotherapy can be administered at discretion of the treating radiation, medical, or gynecologic oncologist. Sequential therapy (radiation followed by chemotherapy) is preferred but not required

Exclusion Criteria:

* Prior abdominal or pelvic irradiation
* Interval between the hysterectomy and planned start of radiotherapy exceeding 16 weeks, unless chemotherapy is administered prior to RT. If chemotherapy is administered prior to RT, consult with PI regarding acceptable time frame.
* Prior history of inflammatory bowel disease
* The diagnosis of another malignancy within =< 2 years before study enrollment, except for those considered to be adequately treated with no evidence of disease or symptoms and/or will not require therapy during the study duration (i.e., basal cell or squamous cell skin cancer, carcinoma in situ of the breast, or bladder or of the cervix)
* Medical, psychiatric, cognitive, or other conditions in the opinion of the investigator that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2027-06-26 (Estimated)

PRIMARY OUTCOMES:
Change in toxicity | Baseline to week 3 of pelvic radiotherapy
  Will be measured with the bowel domain of the Expanded Prostate Cancer Index Composite (EPIC) instrument.
Ability to administer clinical trial to evaluate hypofractionated radiotherapy | Up to 3 years
  Will be measured by percent of eligible patients who begin treatment that complete baseline visit and 3-week EPIC bowel domain questionnaire.

SECONDARY OUTCOMES:
Change in urinary domain of the Expanded Prostate Cancer Index Composite (EPIC) instrument | Baseline to week 3 and 1 year
  estimate impact on acute and 1 year urinary toxicity
Change in gastrointestinal toxicities as collected through Patient-Reported Outcomes instruments (PRO-CTCAE) | Baseline to week 3 and 1 year
  estimate impact upon patient reported gastrointestinal toxicities
Change in Functional Assessment of Cancer Therapy-Cervix (FACT-Cx) | Baseline to week 3 and 1 year
  To assess acute and 1 year quality of life following treatment.
Change in COST-FACIT Measure of Financial Toxicity | Baseline to week 3 and 1 year
  To assess acute and 1 year quality of life following treatment
Decision Regret Scale- summary score | At week 3 and 1 year
  To assess satisfaction with decision-making following treatment.
Overall survival | Time to the earliest of all-cause mortality (event), end of study follow-up (censoring criteria), or loss to follow-up (censoring criteria), assessed up to 3 years
  Will use the Kaplan-Meier method to estimate overall survival throughout three years from the time of completing treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gita Suneja, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No